CLINICAL TRIAL: NCT02572817
Title: A Randomized Double-Blind, Phase 3 Study Comparing the Efficacy and Safety of High-Titer Versus Low-Titer Anti-Influenza Immune Plasma for the Treatment of Severe Influenza A
Brief Title: Comparing the Efficacy and Safety of High-Titer Versus Low-Titer Anti-Influenza Immune Plasma for the Treatment of Severe Influenza A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRC-005; NCT02610478 (obsolete NCT alias)
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Influenza A Virus Infection
Keywords: Anti-Influenza Immune Plasma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-titer anti-influenza plasma (Experimental): Participants received two intravenous infusions of high-titer anti-influenza plasma on Study Day 0.
  Interventions: Biological: High-titer anti-influenza plasma
- Low-titer anti-influenza plasma (Active Comparator): Participants received two intravenous infusions of low-titer anti-influenza plasma on Study Day 0.
  Interventions: Biological: Low-titer anti-influenza plasma

INTERVENTIONS:
Biological: High-titer anti-influenza plasma — Human plasma (FFP or FP24, 225-350 mL per unit or pediatric equivalent) with both an influenza A/H1N1 and A/H3N2 HAI titer of at least 1:80
  Arms: High-titer anti-influenza plasma
Biological: Low-titer anti-influenza plasma — Human plasma (FFP or FP24, 225-350 mL per unit or pediatric equivalent) with both an influenza A/H1N1 and A/H3N2 HAI titer of 1:10 or less
  Arms: Low-titer anti-influenza plasma

SUMMARY:
This study assessed the efficacy and safety of anti-influenza immune plasma, as an addition to standard of care antivirals, in participants hospitalized with severe influenza A infection.

DETAILED DESCRIPTION:
Despite antivirals and vaccines, influenza is responsible for thousands of hospitalizations and deaths each year worldwide. Because of this, additional treatments for influenza are needed. One potential treatment may be the use of high-titer anti-influenza immune plasma. The purpose of this study is to evaluate the efficacy and safety of treatment with high-titer versus low-titer anti-influenza immune plasma, in addition to standard care, in participants hospitalized with severe influenza A infection.

This study enrolled people aged 2 weeks or older who are hospitalized with severe influenza A infection. Participants were randomly assigned to receive either high-titer anti-influenza plasma or low-titer (control) anti-influenza plasma on Day 0. In addition, all participants received standard care antivirals. Participants were assessed on Day 0 (baseline) and on Days 1, 2, 3, 7, 14, and 28. For participants who were not hospitalized on Days 2, 14, and 28, researchers could contact participants by telephone. Study procedures included clinical assessments, blood collection, and oropharyngeal swabs.

ELIGIBILITY:
Inclusion Criteria for Enrollment (Screening):

* Subjects must be aged 2 weeks or older.
* Hospitalization due to signs and symptoms of influenza.

  * Note: The decision for hospitalization will be made by the treating clinician. To be considered eligible, the hospitalization may either be an initial hospitalization, or a prolongation of a hospitalization due to a respiratory illness that was found to be from influenza. Influenza could be a component of a larger respiratory syndrome (i.e. COPD exacerbation thought to be triggered by influenza). However, respiratory syndromes that are not likely due to the virus should not be included (i.e. a subject that had mild influenza then developed pulmonary embolism and respiratory distress from the embolism).
* Study plasma available on-site or available within 24 hours after randomization.
* Not previously screened nor randomized in this study.
* Willingness to have blood and respiratory samples obtained and stored.
* Willingness to return for all required study visits and participate in study follow up.

Inclusion Criteria for Randomization:

* Locally determined positive test for influenza A (by polymerase chain reaction [PCR], other nucleic acid testing, or by rapid Ag) from a specimen obtained less than or equal to 48 hours prior to randomization.
* Onset of illness less than or equal to 6 days before randomization, defined as when the subject first experienced at least one respiratory symptom or fever.
* Note: For subjects with chronic respiratory symptoms (chronic cough, or COPD with baseline dyspnea), the onset of symptoms is defined as the point when the symptoms changed during this illness). Hospitalized due to influenza, with anticipated hospitalization for more than 24 hours after randomization. Criteria for hospitalization will be up to the individual treating clinician.
* National Early Warning (NEW) or Pediatric Early Warning (PEW) score greater than or equal to 3 within 12 hours prior to randomization.
* ABO-compatible plasma available on-site or available within 24 hours after randomization.

Exclusion Criteria for Randomization:

* Strong clinical evidence in the judgment of the site investigator that the etiology of illness is primarily bacterial super-infection in origin. Co-infection would be allowed, as there may be benefit to resolving influenza illness faster. Super-infection, where influenza illness occurred and is resolving, and new bacterial illness causing deterioration should be excluded (e.g., if the subject's respiratory infection is thought unlikely to benefit from additional antiviral therapy, this exclusion criteria would be met).
* Prior treatment with any anti-influenza investigational drug, anti-influenza investigational intravenous immune globulin (IVIG), or anti-influenza investigational plasma therapy within 30 days prior to screening. Other investigational drug therapies (non-influenza) and administration of plasma and/or IVIG for non-influenza reasons are allowed.
* History of allergic reaction to blood or plasma products (as judged by the site investigator).
* A pre-existing condition or use of a medication that, in the opinion of the site investigator, may place the individual at a substantially increased risk of thrombosis (e.g., cryoglobulinemia, severe refractory hypertriglyceridemia, or clinically significant monoclonal gammopathy). Prior IVIG use alone would not meet exclusion criteria, but the investigator should consider the potential for a hyper-coagulable state.
* Subjects who, in the judgment of the site investigator, will be unlikely to comply with the requirements of this protocol, including being not contactable following discharge from hospital.
* Medical conditions for which receipt of 500-600 mL (or pediatric equivalent) of intravenous fluid may be dangerous to the subject (e.g., decompensated congestive heart failure).

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04-26 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beigel, MD, Study Chair — Leidos Biomedical Research, Inc. in support of Clinical Research Section, LIR, NIAID, National Institutes of Health
Locations (30):
- United States (30):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - UCLA Pediatrics Infectious Diseases, Los Angeles, California
  - Naval Medical Center San Diego (NMCSD), San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - University of Florida, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Beaumont Hospital, Troy, Troy, Michigan
  - Mayo Clinic Campus Saint Mary's, Rochester, Minnesota
  - St. Louis Children's Hospital at Washington University, St Louis, Missouri
  - Creighton University Medical Center, Omaha, Nebraska
  - New York University/Bellevue Hospital, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont
  - Madigan Army Medical Center (MAMC), Tacoma, Washington

REFERENCES:
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Leteurtre S, Duhamel A, Grandbastien B, Lacroix J, Leclerc F. Paediatric logistic organ dysfunction (PELOD) score. Lancet. 2006 Mar 18;367(9514):897; author reply 900-2. doi: 10.1016/S0140-6736(06)68371-2. No abstract available. PMID 16546531
- [Background] Leteurtre S, Martinot A, Duhamel A, Proulx F, Grandbastien B, Cotting J, Gottesman R, Joffe A, Pfenninger J, Hubert P, Lacroix J, Leclerc F. Validation of the paediatric logistic organ dysfunction (PELOD) score: prospective, observational, multicentre study. Lancet. 2003 Jul 19;362(9379):192-7. doi: 10.1016/S0140-6736(03)13908-6. PMID 12885479
- [Background] Smith GB, Prytherch DR, Meredith P, Schmidt PE, Featherstone PI. The ability of the National Early Warning Score (NEWS) to discriminate patients at risk of early cardiac arrest, unanticipated intensive care unit admission, and death. Resuscitation. 2013 Apr;84(4):465-70. doi: 10.1016/j.resuscitation.2012.12.016. Epub 2013 Jan 4. PMID 23295778
- [Background] Parshuram CS, Bayliss A, Reimer J, Middaugh K, Blanchard N. Implementing the Bedside Paediatric Early Warning System in a community hospital: A prospective observational study. Paediatr Child Health. 2011 Mar;16(3):e18-22. doi: 10.1093/pch/16.3.e18. PMID 22379384
- [Derived] Beigel JH, Aga E, Elie-Turenne MC, Cho J, Tebas P, Clark CL, Metcalf JP, Ozment C, Raviprakash K, Beeler J, Holley HP Jr, Warner S, Chorley C, Lane HC, Hughes MD, Davey RT Jr; IRC005 Study Team. Anti-influenza immune plasma for the treatment of patients with severe influenza A: a randomised, double-blind, phase 3 trial. Lancet Respir Med. 2019 Nov;7(11):941-950. doi: 10.1016/S2213-2600(19)30199-7. Epub 2019 Sep 30. PMID 31582360

RESULTS

PARTICIPANT FLOW:
Groups:
- High-titer Anti-influenza Plasma mITT: High-titer anti-influenza mITT (modified intent to treat) is the subgroup of high-titer anti-influenza plasma participants who received any study plasma
- Low-titer Anti-influenza Plasma mITT: Low-titer anti-influenza mITT (modified intent to treat) is the subgroup of low-titer anti-influenza plasma participants who received any study plasma
Period: Overall Study
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Started | 91 | 47
Completed | 82 | 41
Not Completed | 9 | 6
Not completed — Death | 6 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT | Total
Number analyzed (Participants) | 91 | 47 | 138
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [47 to 69] | 63 [44 to 69] | 61 [45 to 69]
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 8 | 5 | 13
  ≥ 18 years | 83 | 42 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 26 | 67
  Male | 50 | 21 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2 | 0 | 2
  Asian | 2 | 2 | 4
  Black or African American | 16 | 8 | 24
  White | 69 | 36 | 105
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 91 | 47 | 138
Baseline National Early Warning (NEW) score [Median (Inter-Quartile Range); unit: units on a scale] — The National Early Warning (NEW) score was only measured for the adult participants. The NEW score is used to determine the degree of illness of a patient. Baseline is defined as the Day 0. The NEW score is based on 7 clinical parameters. The total score is reported. The range is from 0 to 20, with lower values representing a better outcome. For more details see protocol section 7.3.2. Population: The NEW score was only measured for the adult participants. Only non-missing scores were summarized.
  units on a scale
    number analyzed (Participants) | 82 | 42 | 124
    (all) | 5 [4 to 8] | 5 [3 to 7] | 5 [4 to 7]
Baseline Pediatric Early Warning (PEW) score [Median (Inter-Quartile Range); unit: units on a scale] — The Pediatric Early Warning (PEW) score was only measured for the pediatric participants. The PEW score is a numerical scoring system to define pediatric patients at risk of clinical deterioration. Baseline is defined as the Day 0. The PEW score is based on 7 clinical parameters. The total score is reported. The range is from 0 to 26, with lower values representing a better outcome. For more details see protocol section 7.3.3. Population: The PEW score was only measured for the pediatric participants.
  units on a scale
    number analyzed (Participants) | 8 | 5 | 13
    (all) | 9 [5 to 11.5] | 8 [4 to 13] | 8 [5 to 12]
Baseline Sequential Organ Failure Assessment (SOFA) Score [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) score was only measured for the adult participants. The SOFA score is a scoring system to determine the extent of a person's organ function or rate of failure. Baseline is defined as the Day 0. The SOFA score is based on six different scores. The total score is reported. The range is from 0 to 24, with lower values representing a better outcome. For more details see protocol section 7.3.4. Population: The SOFA score was only measured for the adult participants. Only non-missing scores were summarized.
  units on a scale
    number analyzed (Participants) | 80 | 41 | 121
    (all) | 3 [1.5 to 6] | 3 [2 to 7] | 3 [2 to 6]
Baseline Pediatric Logistic Organ Dysfunction (PELOD) Score [Median (Inter-Quartile Range); unit: units on a scale] — The Pediatric Logistic Organ Dysfunction (PELOD) score was only measured for the pediatric participants. The PELOD score is an organ dysfunction score that can be used in the pediatric population to sequentially evaluate organ dysfunction and predict mortality. Baseline is defined as the Day 0. The score is based on six different scores. The total score is reported. The range is from 0 to 71, with lower values representing a better outcome. For more details see protocol section 7.3.5. Population: The PELOD score was only measured for the pediatric participants. Only non-missing scores were summarized.
  units on a scale
    number analyzed (Participants) | 8 | 4 | 12
    (all) | 0 [0 to 1] | 3 [1.5 to 12] | 0.5 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status at Day 7
Description: The clinical status at Day 7 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 7
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment (with available data).
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 46
Participants
  Death | 2 | 2
  in ICU | 15 | 10
  Non-ICU hospitalization with supplemental O2 | 16 | 7
  Non-ICU hospitalization without supplemental O2 | 8 | 5
  Not hospitalized, unable for normal activity | 30 | 11
  Not hospitalized, able for normal activity | 20 | 11
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.54, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.65 to 2.29]

2. Secondary Outcome: Clinical Status at Day 1
Description: The clinical status at Day 1 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 1
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 46
Participants
  Death | 0 | 0
  in ICU | 38 | 18
  Non-ICU hospitalization with supplemental O2 | 30 | 14
  Non-ICU hospitalization without supplemental O2 | 21 | 14
  Not hospitalized, unable for normal activity | 2 | 0
  Not hospitalized, able for normal activity | 0 | 0
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.66, Regression, Logistic; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.45 to 1.66]

3. Secondary Outcome: Clinical Status at Day 2
Description: The clinical status at Day 2 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 2
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 46
Participants
  Death | 1 | 0
  in ICU | 35 | 17
  Non-ICU hospitalization with supplemental O2 | 24 | 12
  Non-ICU hospitalization without supplemental O2 | 19 | 13
  Not hospitalized, unable for normal activity | 6 | 3
  Not hospitalized, able for normal activity | 6 | 1
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.87, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.5 to 1.8]

4. Secondary Outcome: Clinical Status at Day 3
Description: The clinical status at Day 3 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 3
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 90 | 43
Participants
  Death | 1 | 0
  in ICU | 29 | 15
  Non-ICU hospitalization with supplemental O2 | 20 | 10
  Non-ICU hospitalization without supplemental O2 | 17 | 12
  Not hospitalized, unable for normal activity | 11 | 4
  Not hospitalized, able for normal activity | 12 | 2
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.49, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.65 to 2.41]

5. Secondary Outcome: Clinical Status at Day 14
Description: The clinical status at Day 14 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 14
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 86 | 45
Participants
  Death | 4 | 4
  in ICU | 10 | 6
  Non-ICU hospitalization with supplemental O2 | 3 | 2
  Non-ICU hospitalization without supplemental O2 | 6 | 1
  Not hospitalized, unable for normal activity | 26 | 12
  Not hospitalized, able for normal activity | 37 | 20
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.83, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.55 to 2.08]

6. Secondary Outcome: Clinical Status at Day 28
Description: The clinical status at Day 28 was based on a 6-point ordinal scale:
  1. Death
  2. In ICU
  3. Non-ICU hospitalization, requiring supplemental oxygen (O2)
  4. Non-ICU hospitalization, not requiring supplemental oxygen
  5. Not hospitalized, but unable to resume normal activities
  6. Not hospitalized with full resumption of normal activities A higher score corresponds to a better health outcome
Time Frame: Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 88 | 45
Participants
  Death | 6 | 4
  in ICU | 5 | 3
  Non-ICU hospitalization with supplemental O2 | 0 | 2
  Non-ICU hospitalization without supplemental O2 | 2 | 1
  Not hospitalized, unable for normal activity | 24 | 11
  Not hospitalized, able for normal activity | 51 | 24
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.47, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.65 to 2.56]

7. Secondary Outcome: Duration of Initial Hospitalization
Description: Duration (in days) of initial hospitalization, restricted to duration between randomization and last visit
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
days | 5 [3 to 12] | 6 [4 to 12]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.3, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: 28-day Mortality
Description: Number of deaths during study follow-up
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants | 6 | 4
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.64, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.21 to 2.64]

9. Secondary Outcome: In-hospital Mortality During Initial Hospitalization
Description: Number of deaths in the hospital during initial hospitalization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants | 4 | 3
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.69, Fisher Exact

10. Secondary Outcome: Composite of Mortality and Hospitalization at Day 7, Day 14, Day 28
Description: Two categories were considered for the composite of mortality and hospitalization:
  Dead or hospitalized Alive and not hospitalized
Time Frame: Day 7, Day 14, Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants
  Composite mortality and hospitalization, Day 7: number analyzed (Participants) | 91 | 46
  Composite mortality and hospitalization, Day 7: Dead or hospitalized | 41 | 24
  Composite mortality and hospitalization, Day 7: Alive and not hospitalized | 50 | 22
  Composite mortality and hospitalization, Day 14: number analyzed (Participants) | 86 | 45
  Composite mortality and hospitalization, Day 14: Dead or hospitalized | 23 | 13
  Composite mortality and hospitalization, Day 14: Alive and not hospitalized | 63 | 32
  Composite mortality and hospitalization, Day 28: number analyzed (Participants) | 88 | 45
  Composite mortality and hospitalization, Day 28: Dead or hospitalized | 13 | 10
  Composite mortality and hospitalization, Day 28: Alive and not hospitalized | 75 | 35
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Composite mortality and hospitalization, Day 7; Test type: Superiority; p = 0.43, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.65 to 2.71]
Statistical Analysis 2: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Composite mortality and hospitalization, Day 14; Test type: Superiority; p = 0.79, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.5 to 2.48]
Statistical Analysis 3: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Composite mortality and hospitalization, Day 28; Test type: Superiority; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [0.66 to 4.12]

11. Secondary Outcome: Change From Baseline to Day 3 and Day 7 in National Early Warning (NEW) Score
Description: The National Early Warning (NEW) score was only measured for the adult participants.
  The range of the NEW score is from 0 to 20, with lower values representing a better outcome.
  Baseline is defined as the Day 0. Change was defined as the value at Day 3 or Day 7 minus the value at baseline.
Time Frame: Day 0, Day 3, Day 7
Population: Modified intent-to-treat adult population: subgroup of randomized adult participants who received any study treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 83 | 42
units on a scale
  Change in NEW from baseline to Day 3: number analyzed (Participants) | 77 | 42
  Change in NEW from baseline to Day 3 | -2 [-4 to 0] | -1 [-3 to 0]
  Change in NEW from baseline to Day 7 | -2 [-4 to 0] | -2 [-4 to -0.5]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in NEW from baseline to Day 3; Test type: Superiority; p = 0.2, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = -1, 95% CI 2-sided [-2 to 0]
Statistical Analysis 2: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in NEW from baseline to Day 3; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = 0, 95% CI 2-sided [-1 to 1]

12. Secondary Outcome: Change From Baseline to Day 3 and Day 7 in Pediatric Early Warning (PEW) Score
Description: The Pediatric Early Warning (PEW) score was only measured for the pediatric participants.
  The range is from 0 to 26, with lower values representing a better outcome. Baseline is defined as the Day 0. Change was defined as the value at Day 3 or Day 7 minus the value at baseline.
Time Frame: Day 0, Day 3, Day 7
Population: Modified intent-to-treat pediatric population: subgroup of randomized pediatric participants who received any study treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 8 | 5
units on a scale
  Change in PEW from baseline to Day 3 | 0 [-3 to 2] | -1 [-6 to -1]
  Change in PEW from baseline to Day 7 | -4.5 [-7 to -0.5] | -5 [-8 to -3]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in PEW from baseline to Day 3; Test type: Superiority; p = 0.18, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in PEW from baseline to Day 7; Test type: Superiority; p = 0.61, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Duration of Supplemental Oxygen
Description: Duration (in days) of total supplemental oxygen use among those participants who required new or increased oxygen at randomization.
  The duration is restricted to duration between randomization and last visit.
Time Frame: From Day 0 to Day 28 visit. The window of the Day 28 visit was 28-32 days from study entry.
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who required new or increased oxygen at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 65 | 34
days | 6 [3 to 21] | 7 [3 to 29]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = 0, 95% CI 2-sided [-2 to 1]

14. Secondary Outcome: Incidence of New Oxygen Use During the Study
Description: Incidence of new oxygen use during the study among those participants who did not require oxygen at randomization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who did not require oxygen at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 20 | 11
Participants
  Yes | 7 | 3
  No | 13 | 8
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.98, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [0.23 to 11.01]

15. Secondary Outcome: Duration of Intensive Care Unit (ICU) Stay
Description: Duration (in days) of ICU stay among those participants who were in ICU at randomization.
  The duration is restricted to duration between randomization and last visit.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were in the ICU at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 40 | 20
days | 5 [3.5 to 12.5] | 8 [4 to 25]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = -1.5, 95% CI 2-sided [-6 to 2]

16. Secondary Outcome: Incidence of New ICU Admission Use During the Study
Description: Incidence of new ICU admission during the study among those participants who were not in ICU at randomization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were not in the ICU at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 51 | 27
Participants
  Yes | 3 | 0
  No | 48 | 27
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.55, Fisher Exact

17. Secondary Outcome: Duration of Mechanical Ventilation Use
Description: Duration (in days) of mechanical ventilation use among those participants who were on mechanical ventilation at randomization.
  The duration is restricted to duration between randomization and last visit.
Time Frame: From Day 0 to Day 28 visit. The window of the Day 28 visit was 28-32 days from study entry
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were on mechanical ventilation at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 25 | 14
days | 9 [4 to 16] | 15.5 [7 to 29]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = -3, 95% CI 2-sided [-14 to 2]

18. Secondary Outcome: Incidence of New Mechanical Ventilation Use Stay Use During the Study
Description: Incidence of new mechanical ventilation use during the study among those participants who were not on mechanical ventilation at randomization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were not on mechanical ventilation at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 66 | 33
Participants
  Yes | 3 | 2
  No | 63 | 31
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 1, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.08 to 9.29]

19. Secondary Outcome: Duration of Acute Respiratory Distress Syndrome (ARDS)
Description: Duration (in days) of ARDS use among those participants with ARDS at randomization.
  The duration is restricted to duration between randomization and last visit.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants with ARDS at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 15 | 3
days | 9 [4 to 15] | 8 [4 to 29]

20. Secondary Outcome: Incidence of New ARDS During the Study
Description: Incidence of new ARDS during the study among those participants without ARDS at randomization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants without ARDS at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 75 | 44
Participants
  Yes | 3 | 5
  No | 72 | 39
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.24, Regression, Logistic; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.05 to 1.79]

21. Secondary Outcome: Duration of Extracorporeal Membrane Oxygenation (ECMO)
Description: Duration (in days) of ECMO use among those participants on ECMO at randomization.
  The duration is restricted to duration between randomization and last visit.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were on ECMO at randomization.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 5 | 1
days | 16 [14 to 18] | 20 [20 to 20]

22. Secondary Outcome: Incidence of New ECMO Use During the Study
Description: Incidence of new ECMO use during the study among those participants not on ECMO at randomization
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment, further subset to those participants who were not on ECMO at randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 86 | 46
Participants
  Yes | 1 | 0
  No | 85 | 46
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 1, Fisher Exact

23. Secondary Outcome: Change From Baseline to Day 3 and Day 7 in Sequential Organ Failure Assessment (SOFA) Score
Description: The Sequential Organ Failure Assessment (SOFA) score was only measured for the adult participants.
  The range is from 0 to 24, with lower values representing a better outcome. Baseline is defined as the Day 0. Change was defined as the value at Day 3 or Day 7 minus the value at baseline.
Time Frame: Day 0, Day 3, Day 7
Population: Modified intent-to-treat adult population: subgroup of randomized adult participants who received any study treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 75 | 40
units on a scale
  Change in SOFA from baseline to Day 3 | 0 [-1 to 0] | 0 [-1 to 0]
  Change in SOFA from baseline to Day 7 | -1 [-2 to 0] | 0 [-2 to 1]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in SOFA from baseline to Day 3; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = 0, 95% CI 2-sided [-1 to 0]
Statistical Analysis 2: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in SOFA from baseline to Day 7; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney); Hodges-Lehman estimate of location shift = -1, 95% CI 2-sided [-1 to 0]

24. Secondary Outcome: Change From Baseline to Day 3 and Day 7 in Pediatric Logistic Organ Dysfunction (PELOD) Score
Description: The Pediatric Logistic Organ Dysfunction (PELOD) score was only measured for the pediatric participants.
  The range is from 0 to 71, with lower values representing a better outcome. Baseline is defined as the Day 0. Change was defined as the value at Day 3 or Day 7 minus the value at baseline.
Time Frame: Day 0, Day 3, Day 7
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 8 | 4
units on a scale
  Change in PELOD from baseline to Day 3 | 0 [0 to 9.5] | 10 [5 to 14]
  Change in PELOD from baseline to Day 7 | 0 [0 to 4.5] | 0 [-1.5 to 0]
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in PELOD from baseline to Day 3; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Change in PELOD from baseline to Day 7; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)

25. Secondary Outcome: Disposition After Initial Hospitalization
Description: Disposition at discharge after initial hospitalization was categorized as follows:
  Death, Ongoing at 28 days, Chronic nursing facility, Rehabilitation, Home with home health care, Home without assistance.
  The number of deaths at discharge after initial hospitalization do not necessarily match the overall number of deaths.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants
  Death | 4 | 4
  Ongoing at 28 days | 3 | 3
  Chronic nursing facility/ | 7 | 4
  Rehabilitation | 4 | 3
  Home with home health care | 13 | 8
  Home without assistance | 60 | 25
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.12, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.87 to 3.44]

26. Secondary Outcome: Detectable Influenza Virus at Day 3
Description: Detectable influenza virus at Day 3 in oropharyngeal samples
Time Frame: Day 3
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment. This group was further subset wo those with available OP sample results at Day 3.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 85 | 40
Participants
  Detectable | 65 | 35
  Undetectable | 20 | 5
Statistical Analysis 1: Comparison: High-titer Anti-influenza Plasma mITT vs Low-titer Anti-influenza Plasma mITT; Test type: Superiority; p = 0.23, Regression, Logistic; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.13 to 1.43]

27. Secondary Outcome: Hemagglutination Inhibition Assay (HAI) Titers at Days 1, 3, 7 for A/H1N1
Description: Hemagglutination inhibition assay (HAI) titers as measured by serial dilutions at Days 1, 3, 7 for A/H1N1. HAI for A/H1N1 was tested in all influenza seasons while the study was ongoing.
Time Frame: Day 1, Day 3, Day 7
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Geometric Mean (95% Confidence Interval); unit: ratios
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
ratios
  Day 1: number analyzed (Participants) | 87 | 43
  Day 1 | 46.9 [38.5 to 57.1] | 19.7 [13.9 to 27.8]
  Day 3: number analyzed (Participants) | 87 | 41
  Day 3 | 50.6 [40.9 to 62.6] | 23.7 [16.7 to 33.6]
  Day 7: number analyzed (Participants) | 82 | 37
  Day 7 | 63.1 [49.5 to 80.6] | 37.1 [23.2 to 59.4]

28. Secondary Outcome: Hemagglutination Inhibition Assay (HAI) Titers at Days 1, 3, 7 for A/HongKong/4801/2014 H3N2
Description: Hemagglutination inhibition assay (HAI) titers as measured by serial dilutions at Days 1, 3, 7 for A/HongKong/4801/2014 H3N2. HAI for A/HongKong/4801/2014 H3N2 was tested in all influenza seasons while the study was ongoing.
Time Frame: Day 1, Day 3, Day 7
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment
Measure: Geometric Mean (95% Confidence Interval); unit: ratios
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
ratios
  Day 1: number analyzed (Participants) | 87 | 43
  Day 1 | 53.7 [43.2 to 66.7] | 22.4 [16.6 to 30.3]
  Day 3: number analyzed (Participants) | 87 | 41
  Day 3 | 55.2 [44 to 69.4] | 36.8 [24.6 to 36.8]
  Day 7: number analyzed (Participants) | 82 | 37
  Day 7 | 75.7 [57.5 to 99.8] | 53 [30.9 to 90.7]

29. Secondary Outcome: Number of Participants With Grade 3 and 4 Adverse Events (AEs).
Description: Number of participants with reported grade 3 and 4 adverse events (AEs) throughout the study duration. In cases where participants had multiple reports of grade 3 and 4 AEs, they were only counted once.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants | 34 | 14

30. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs).
Description: Number of participants with reported serious adverse events (SAEs) throughout the study duration.
Time Frame: From Day 0 to Day 28
Population: Modified intent-to-treat population: subgroup of randomized participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
Number analyzed (Participants) | 91 | 47
Participants | 31 | 15

ADVERSE EVENTS:
Time Frame: From study entry (Day 0) to Day 28
Description: The protocol required reporting of all grade 3 and 4 adverse events (AEs), all serious AEs and any AE leading to plasma discontinuation (regardless of grade). Clinically evident diagnoses were recorded as AEs. All worsening laboratory values were evaluated as potential AEs. The grading reference was the "Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events" Version 2.0, November 2014.
Arm/Group | High-titer Anti-influenza Plasma mITT | Low-titer Anti-influenza Plasma mITT
All-Cause Mortality (participants affected / at risk) | 6/91 | 4/47
Serious Adverse Events (participants affected / at risk) | 31/91 | 15/47
Other Adverse Events (participants affected / at risk) | 0/91 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-titer Anti-influenza Plasma mITT (N=91) | Low-titer Anti-influenza Plasma mITT (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT02572817/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT02572817/SAP_001.pdf